CLINICAL TRIAL: NCT00857753
Title: A Study to Evaluate the Relative Bioavailability of a Fentanyl PAtch Transdermal Delivery System (25 ug/hr) (Sandoz) Compared to Duragesic (Fentanyl Transdermal SYstem 25 ug/hr Patches (Alza)
Brief Title: Relative Bioavailability of a Fentanyl Patch
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D., VP Product Development, Sandoz, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10613401
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2009-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Fentanyl

ARMS (2):
- 1 (Experimental): Fentanyl patch 25 ug/hr Sandoz
  Interventions: Drug: Fentanyl patch 25 ug/nr Sandoz
- 2 (Active Comparator): Duragesic Patch 25 ug/hr
  Interventions: Drug: Duragesic

INTERVENTIONS:
Drug: Fentanyl patch 25 ug/nr Sandoz
  Arms: 1
Drug: Duragesic
  Arms: 2

SUMMARY:
Tohe purpose of this study is to demonstrate the bioequivalence of a fentanyl patch transdermal delivery system.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on physical exam, medical history or clinical laboratory tests on screening.

Exclusion Criteria:

* Negative test for HIV and hepatitis B and C
* No history of drug or alcohol treatment
* No allergies to opiates

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2006-09; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence according to US FDA guidelines | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Darin B. Brimhall, D.O., Principal Investigator — Novum Pharmaceutical Research Services